CLINICAL TRIAL: NCT03413527
Title: Examining the Impact of Transcranial Magnetic Stimulation (rTMS) on Schizophrenia and Related Disorders: A Case Series
Brief Title: rTMS Treatment for Positive and Negative Symptoms of Schizophrenia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Gary Chaimowitz, Principal Investigator, Head of Forensics Service, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3864
Record Dates: First submitted 2018-01-17; First posted 2018-01-29 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia
Keywords: rTMS
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rTMS Treatment (Experimental)
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — rTMS Treatment

SUMMARY:
This study will examine the effects of rTMS on the negative and positive symptoms of schizophrenia using 2 treatments in sequence applied to related brain areas.

ELIGIBILITY:
Inclusion Criteria:

1. are voluntary and competent to consent to treatment
2. have a diagnosis of schizophrenia or schizoaffective disorder
3. are between the ages of 18 and 75
4. are willing and able to adhere to the treatment schedule
5. Pass the TMS adult safety-screening (TASS) questionnaire
6. have normal thyroid functioning based on pre-study blood work. Patients may be reassessed for the study once thyroid levels have normalized.
7. are willing and able to cooperate with interviews and follow simple instructions

Exclusion Criteria:

1. do not pass the TASS Safety Screening Questionnaire
2. have a significant history of seizures
3. have active suicidal intent
4. are pregnant or may be pregnant. A pregnancy test will be performed for fertile women.
5. have failed a course of Electroconvulsive Therapy (ECT) in the current or previous episode
6. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, or head trauma resulting in loss of consciousness greater than or equal to 5 minutes
7. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
8. have had changes in dose or initiation of any psychotropic medication in the 4 weeks prior to screening. Patients may be re-screened once medications have been stable for 4 weeks.
9. currently (or in the last 4 weeks) take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale (PANSS) | Change from pre-treatment to post treatment over 6 weeks
  semi-structured interview designed to rate the severity of schizophrenia symptoms. Score from 0-231, with higher score being worse.

SECONDARY OUTCOMES:
Beck Depression Inventory | Change from pre-treatment to post treatment over 6 weeks
  Self-report questionnaire for depression symptoms. Scores range from 0-63, with higher being worse.
Hamilton Depression Rating Scale (HAM-D) | change from pre-treatment to post treatment over 6 weeks
  Clinician-rated scale for depression symptoms. Scores range from 0-53, with higher being worse.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Chaimowitz, MD, FRCPC, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No